CLINICAL TRIAL: NCT01747837
Title: REnal SympathetiC Denervation to sUpprEss Tachyarrhythmias in ICD Recipients
Acronym: RESCUE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vivek Reddy (Other)
Responsible Party: Sponsor-Investigator, Vivek Reddy, Director Cardiac Arrhythmia Service, Professor of Medicine, Icahn School of Medicine at Mount Sinai
Organization: Icahn School of Medicine at Mount Sinai (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 12-02-213
Record Dates: First submitted 2012-11-01; First posted 2012-12-12 (Estimated); Results first posted 2020-01-27 (Actual); Last update posted 2020-03-04 (Actual); Status verified 2020-02

CONDITIONS: Ventricular Tachycardia
Keywords: Renal sympathetic denervation; Renal catheter ablation; Ventricular tachycardia
MeSH Terms: conditions — Tachycardia, Ventricular | interventions — Denervation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- standard ICD implantation alone (No Intervention): These subjects will undergo standard ICD implantation alone (if not already present)
- Boston Scientific Vessix Renal Denervation System (Experimental): These subjects will undergo standard ICD implantation (if not already present) plus renal sympathetic denervation.
  Ablation arm
  Interventions: Device: Boston Scientific Vessix Renal Denervation System

INTERVENTIONS:
Device: Boston Scientific Vessix Renal Denervation System — Renal sympathetic denervation is modulation of the nerves which run along the renal arteries (the renal sympathetic nerves) with radiofrequency energy. This is the same energy source used to perform your heart ablation.
  Boston Scientific Vessix Renal Denervation System, Boston Scientific, Inc., Quincy, Massachusetts
  Other Names: Renal sympathetic denervation; Renal denervation; Denervation
  Arms: Boston Scientific Vessix Renal Denervation System

SUMMARY:
The objective of this trial is to determine the efficacy and safety of adjunctive catheter-based renal sympathetic denervation (RSDN) in the primary prevention of implantable cardioverter defibrillator (ICD) therapy in patients with ischemic or non-ischemic ventricular dysfunction, who are to receive an ICD for either i) secondary prevention, or ii) primary prevention + inducible ventricular tachycardia (VT) by programmed ventricular stimulation at the time of ICD implantation. These patients will be randomized to ICD alone or ICD + RSDN.

DETAILED DESCRIPTION:
Rationale for this Study

Despite significant advances in the management of ventricular arrhythmias through the use of ICD therapy, anti-arrhythmic drugs (AADs), and catheter-based ablation strategies, considerable challenges remain. The optimal method for the prevention of ICD shocks remains unclear. RSDN may be an effective tool for preventing ventricular arrhythmias, and associated ICD therapies, by reducing central sympathetic tone, catecholamine levels, and the renin-angiotensin-aldosterone system. Although RSDN has been shown to reduce the recurrence of VT in a case report of 2 patients suffering from electrical storm, to date no large prospective randomized study has evaluated the impact of RSDN in the primary prevention of ICD therapy in patients with ischemic or non-ischemic ventricular dysfunction. Also of note, there is data suggesting that RSDN may even decrease the rate of supraventricular arrhythmias such as atrial fibrillation. Thus, RESCUE will specifically evaluate the safety and efficacy of RSDN in the prevention of ICD therapy in patients with ventricular dysfunction who are to receive an ICD for either secondary prevention, or primary prevention if they have inducible VT by programmed ventricular stimulation at the time of ICD implantation.

Description of Procedures

Screening:

To take part in this study, you must meet all study requirements. The screening visit tests and procedures are done to see if you are eligible to be in the study. The study doctor will review these with you and let you know if you qualify. The study doctor will make a final decision about your possible study qualification.

Pre-randomization Procedures:

After providing written consent the following data will be collected and examinations and tests performed:

* A physical examination
* Your blood pressure will be taken
* A review of your medical history and what medications you are taking
* A blood sample will be drawn for routine laboratory tests.
* Women who can have children will take a urine pregnancy test. The test must be negative for you to be in this study.
* A Transthoracic Echocardiogram (TTE)-a non-invasive test where a probe is placed on the chest wall and images are taken through the chest wall of the heart valves and heart muscle, that will measure the left ventricular size (heart wall thickness) and mitral inflow (flow of blood through the heart valve).
* An ICD interrogation (if you already have an ICD implanted) - a non-invasive test where a device is placed over the chest wall near your ICD, and data is transmitted wirelessly from your ICD to a laptop for your physician to review.
* An electrocardiogram (EKG) - a non-invasive test where several probes are placed on the chest wall that will measure electrical activity in your heart.

Randomization:

Immediately following the catheter ablation, patients will undergo a renal angiogram in order to assess suitability for catheter-based renal sympathetic denervation. A renal angiogram is an x-ray study of the blood vessels in the kidney to evaluate for blockage, and abnormalities that could be affecting the blood supply to the kidney. It is performed by injecting contrast dye through a catheter (a tiny tube) into the blood vessels of the kidney. The study doctor will assess whether the renal arteries are suitable to receive catheter-based renal denervation. Once you agree to participate in this study, by signing this informed consent, and are it is determined that you are eligible to participate you will be randomized to one of two treatment groups immediately following the renal angiogram.

Randomization means that you are put into a group by chance. It is like flipping a coin. You will have an equal chance (50%) of being placed in either group. This study design is single-blinded; you will not know ahead of time which group you will be in. Only your physician will know which group you are randomized to.

If you do not already have an ICD, you will undergo ICD placement as part of routine clinical care. You may undergo ICD placement up to 1 month (30 days) before randomization. An ICD (implantable cardioverter-defibrillator) is a small battery-powered electrical impulse generator which is implanted in patients who are at risk of sudden cardiac death due to ventricular fibrillation and ventricular tachycardia. The device is programmed to detect abnormal heart beats (cardiac arrhythmia) and correct it by delivering a jolt of electricity.

The first group will undergo catheter-based sympathetic renal denervation. Renal Sympathetic Denervation is a procedure that uses a catheter probe inserted into the renal (kidney) artery that deactivates the nerves that are linked to high blood pressure.

The second group (control group) will receive no further intervention after ICD implantation.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 years of age
* Structural heart disease (post-MI, dilated cardiomyopathy, sarcoid myopathy, hypertrophic cardiomyopathy, etc.)
* Planned for ICD implantation for:

  * i. Secondary prevention (eg: VT/VF arrest, sustained VT, syncope/inducible VT)
  * ii. Primary prevention + inducible MMVT during induction via ICD lead testing
* Accessibility of renal vasculature (determined by renal angiography)
* Ability to understand the requirements of the study
* Willingness to adhere to study restrictions and comply with all post- procedural follow-up requirements

Exclusion Criteria:

* Patient taking a Class I or III antiarrhythmic drug.
* Planned to undergo a cardiac VT ablation procedure
* NYHA Class IV Congestive Heart Failure
* MI within 30 days
* Known renovascular abnormalities that would preclude RSDN (eg, renal artery stenosis, previous renal artery stenting or angioplasty)
* Baseline orthostatic hypotension
* End stage renal failure on dialysis
* Life expectancy <1 year for any medical condition
* Known pregnancy or positive β-HCG within 7 days of procedure.
* Coronary Artery Bypass Graft (CABG) within 30 days of the procedure

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2015-10-22 (Actual); Primary Completion 2019-01-09 (Actual); Study Completion 2019-01-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Vivek Reddy, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (4):
- United States (2):
  - Mount Sinai Hospital, New York, New York
  - Texas Cardiac, Austin, Texas
- Na Homolce Hospital, Prague, Czechia
- Academician E.N. Meshalkin Novosibirsk State Budget Research Institute of Circulation Pathology, Novosibirsk, Russia

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: First enrollment on Oct 22, 2015.
  Last enrollment on May 3, 2017 with last study visit date conducted on Jan 9, 2019,
  50 participants consented, 2 were found ineligible due to irregular renal anatomy during the angiography and not randomized.
Groups:
- Boston Scientific Vessix Renal Denervation System: These subjects will undergo standard ICD implantation (if not already present) plus renal sympathetic denervation.
  Boston Scientific Vessix Renal Denervation System: Renal sympathetic denervation is modulation of the nerves which run along the renal arteries (the renal sympathetic nerves) with radiofrequency energy. This is the same energy source used to perform your heart ablation.
  Boston Scientific Vessix Renal Denervation System, Boston Scientific, Inc., Quincy, Massachusetts
Period: Overall Study
Arm/Group | Standard ICD Implantation Alone | Boston Scientific Vessix Renal Denervation System
Started | 25 | 23
Completed | 16 | 17
Not Completed | 9 | 6
Not completed — Lost to Follow-up | 5 | 2
Not completed — Death | 4 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard ICD Implantation Alone | Boston Scientific Vessix Renal Denervation System | Total
Number analyzed (Participants) | 25 | 23 | 48
Age, Continuous [Mean (Standard Deviation); unit: years] | 64 (10.76) | 63.3 (10.82) | 63.7 (10.68)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 3 | 9
  Male | 19 | 20 | 39
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 24 | 23 | 47
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 2 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 24 | 21 | 45
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Time to First Event Requiring ICD Therapy or Incessant VT
Description: The primary endpoint of this study is the time to first event requiring implantable cardioverter defibrillator (ICD) therapy or Incessant VT. (Ventricular tachycardia (VT) occurring below the ICD rate cut-off); this will be assessed in the on-treatment patient cohort. An event requiring ICD therapy is defined as an anti-tachycardia pacing (ATP) or shock therapy for ventricular tachycardia or fibrillation.
Time Frame: 24 months
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Standard ICD Implantation Alone | Boston Scientific Vessix Renal Denervation System
Number analyzed (Participants) | 25 | 23
days | 177.2 (148.65) | 148.66 (148.6)

2. Secondary Outcome: Number of Occurrences of Appropriate ICD Therapy
Description: Number of Occurrences of Appropriate ICD therapy assessed in the full intention-to-treat patient cohort. An Appropriate ICD therapy is defined as anti-tachycardia pacing (ATP) or shock therapy for ventricular tachycardia or fibrillation.
Time Frame: 24 months
Measure: Mean (Standard Deviation); unit: Occurences
Arm/Group | Standard ICD Implantation Alone | Boston Scientific Vessix Renal Denervation System
Number analyzed (Participants) | 25 | 23
Occurences | 46 (3.78) | 122 (20.2)

3. Secondary Outcome: Number of Occurrences of Inappropriate ICD Therapy
Description: Number of occurrences of inappropriate shocks. Inappropriate ICD therapy are shocks given by the ICD for atrial fibrillation, supraventricular tachycardia or an abnormal sensing.
Time Frame: 24 months
Measure: Mean (Standard Deviation); unit: Occurrences
Arm/Group | Standard ICD Implantation Alone | Boston Scientific Vessix Renal Denervation System
Number analyzed (Participants) | 25 | 23
Occurrences | 388 (70.4) | 86 (15.8)

4. Secondary Outcome: Number of Hospitalizations for Cardiovascular Causes
Description: Cumulative number of Hospitalizations for Cardiovascular Causes
Time Frame: 24 months
Population: cumulative number of hospitalizations
Measure: Number; unit: hospitalizations
Arm/Group | Standard ICD Implantation Alone | Boston Scientific Vessix Renal Denervation System
Number analyzed (Participants) | 25 | 23
hospitalizations | 11 | 9

5. Secondary Outcome: Number of Episodes of Total VT Burden
Description: Cumulative Number of episodes of Total VT burden
Time Frame: 24 months
Measure: Number; unit: Episodes
Arm/Group | Standard ICD Implantation Alone | Boston Scientific Vessix Renal Denervation System
Number analyzed (Participants) | 25 | 23
Episodes | 513 | 671

6. Secondary Outcome: All-Cause Mortality
Description: All-Cause Mortality
Time Frame: 24 months
Measure: Count of Participants; unit: Participants
Arm/Group | Standard ICD Implantation Alone | Boston Scientific Vessix Renal Denervation System
Number analyzed (Participants) | 25 | 23
Participants | 4 | 4

7. Secondary Outcome: Number of Occurrence of ICD Storm
Description: The cumulative number of occurrences of ICD storm, defined as ≥3 appropriate shock therapies within 24 hours
Time Frame: 24 months
Measure: Number; unit: occurences
Arm/Group | Standard ICD Implantation Alone | Boston Scientific Vessix Renal Denervation System
Number analyzed (Participants) | 25 | 23
occurences | 1 | 2

8. Secondary Outcome: BUN Measurements
Description: Blood Urea Nitrogen (BUN) measurements
Time Frame: baseline, 6 months, 12 months, 24 months
Population: data only available for those participants who returned for respective study visits
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Standard ICD Implantation Alone | Boston Scientific Vessix Renal Denervation System
Number analyzed (Participants) | 25 | 23
mmol/L
  Baseline | 13.31 (6.24) | 10.6 (4.33)
  6 months: number analyzed (Participants) | 23 | 20
  6 months | 12 (5.77) | 11.71 (7.45)
  12 months: number analyzed (Participants) | 20 | 19
  12 months | 10.02 (5.76) | 8.71 (6.87)
  24 months: number analyzed (Participants) | 13 | 12
  24 months | 9.09 (3.75) | 8 (3.31)

9. Secondary Outcome: Creatinine Measurements
Description: Creatinine measurements
Time Frame: baseline, 6 months, 12 months, 24 months
Population: data only available for those participants who returned for respective study visits
Measure: Mean (Standard Deviation); unit: µmol/L
Arm/Group | Standard ICD Implantation Alone | Boston Scientific Vessix Renal Denervation System
Number analyzed (Participants) | 25 | 23
µmol/L
  Baseline | 105 (32.57) | 102 (20.68)
  6 months: number analyzed (Participants) | 23 | 20
  6 months | 108 (24.6) | 108 (43.12)
  12 months: number analyzed (Participants) | 20 | 19
  12 months | 110 (35.28) | 104 (28.6)
  24 months: number analyzed (Participants) | 13 | 12
  24 months | 107 (24.97) | 98 (14.24)

10. Secondary Outcome: Procedure Related Adverse Events
Description: Procedure related adverse events including, but not limited to hematomas, pseudoaneurysms and renal artery stenosis.
Time Frame: 24 months
Measure: Number; unit: Events
Arm/Group | Standard ICD Implantation Alone | Boston Scientific Vessix Renal Denervation System
Number analyzed (Participants) | 25 | 23
Events | 2 | 7

11. Secondary Outcome: Number of Participants With Orthostatic Hypotension
Description: Number of participants who developed of orthostatic hypotension
Time Frame: 24 months
Measure: Count of Participants; unit: Participants
Arm/Group | Standard ICD Implantation Alone | Boston Scientific Vessix Renal Denervation System
Number analyzed (Participants) | 25 | 23
Participants | 0 | 0

12. Secondary Outcome: Number of Participants With Major Complication
Description: Number of Participants with Major Complication defined as death, stroke, myocardial infarction (MI) or any other serious adverse events related to the treatment or procedure within the first 30 days or through hospital discharge (whichever is longer)
Time Frame: average 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | Standard ICD Implantation Alone | Boston Scientific Vessix Renal Denervation System
Number analyzed (Participants) | 25 | 23
Participants | 0 | 3

ADVERSE EVENTS:
Time Frame: 24 months
Arm/Group | Standard ICD Implantation Alone | Boston Scientific Vessix Renal Denervation System
All-Cause Mortality (participants affected / at risk) | 4/25 | 4/23
Serious Adverse Events (participants affected / at risk) | 10/25 | 11/23
Other Adverse Events (participants affected / at risk) | 3/25 | 6/23
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Standard ICD Implantation Alone (N=25) | Boston Scientific Vessix Renal Denervation System (N=23)
Anemia (Blood and lymphatic system disorders) | 0 | 1
Bedsore of pocket ICD (Infections and infestations) | 0 | 1
Cardiac Arrhythmias (Cardiac disorders) | 3 | 2
Collapse (General disorders) | 1 | 1
Dyspepsia (Gastrointestinal disorders) | 0 | 1
Emphysema Thoracalgia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Episode of Chest Pain (Cardiac disorders) | 0 | 1
Heart Failure (Cardiac disorders) | 4 | 1
Hip Fracture (Musculoskeletal and connective tissue disorders) | 1 | 0
Hip Surgery (Musculoskeletal and connective tissue disorders) | 0 | 1
Implantation of BIV IC (Surgical and medical procedures) | 1 | 0
Ischemic Stroke (General disorders) | 1 | 0
Myocardial Infarction (Cardiac disorders) | 0 | 2
Pleural Effusion (Cardiac disorders) | 1 | 0
Pocket Hematoma (Skin and subcutaneous tissue disorders) | 1 | 1
Pocket Revision (Surgical and medical procedures) | 0 | 1
Skin erosion on the place of ICD (Infections and infestations) | 1 | 0
Stable exertional angina (Cardiac disorders) | 1 | 1
Syncope (General disorders) | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Standard ICD Implantation Alone (N=25) | Boston Scientific Vessix Renal Denervation System (N=23)
Acute Respiratory Infection (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dislocation of the Atrial Electrode (Surgical and medical procedures) | 0 | 1
Groin Hematoma (Skin and subcutaneous tissue disorders) | 0 | 1
Neoplasm of Left Kidney (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Puncture (Cardiac disorders) | 1 | 0
Renal Artery Stenosis (Renal and urinary disorders) | 0 | 2
Cardiac Arrhythmias (Cardiac disorders) | 1 | 0
Collapse (General disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-10-20): https://cdn.clinicaltrials.gov/large-docs/37/NCT01747837/Prot_SAP_000.pdf